CLINICAL TRIAL: NCT04710095
Title: Perceived Alcohol Reward Value and Risk: Neural Correlates and Treatment Effects
Brief Title: Perceived Alcohol Rewards and Risks Study
Acronym: PARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, PhD, Co-Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#15-000237; R21AA023669 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Heavy Drinking
MeSH Terms: interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Alcohol Intervention (Active Comparator): A brief intervention consisting of a 30-45 minute individual face-to-face session based on the principles of motivational interviewing.
  Interventions: Behavioral: Brief Alcohol Intervention
- Attention-Matched Control Condition (Sham Comparator): Brief attention-matched control condition.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention — Brief alcohol intervention uses a motivational interviewing approach and covers the following components: giving information about the possible health risks associated with alcohol use, placing the responsibility for change on the individual, discussing the reasons for drinking and downsides of drinking, and setting a goal and change plan if the participant is receptive.
  Arms: Brief Alcohol Intervention
Behavioral: Control Condition — The attention-matched control condition consisting of a 30-min video about astronomy.
  Arms: Attention-Matched Control Condition

SUMMARY:
The identification of mechanisms that underlie how people reduce or eliminate alcohol use is a critical public health issue. Understanding these mechanisms can inform how to effectively intervene with problem drinkers. Thus far it has been a challenge for the alcohol research field to find consistent empirical evidence in support of candidate mechanisms of behavior change. Scientific advancement in this area may be aided by longitudinal transdisciplinary research on the interplay between behavioral intervention, cognition, and brain activity to understand underlying processes of behavior change among heavy drinkers. This study employed a randomized 2-arm repeated measures design with a sample of non-treatment seeking adult heavy drinkers to examine changes in perceived reward value and risks of alcohol use as a mechanism of alcohol behavior change after a brief behavioral intervention. Participants were randomized to either a 1-session behavioral intervention or to an attention-matched control condition and immediately after completed an fMRI scan. The focus of this project is to examine if group differences in perceived alcohol reward value after the intervention mediates an intervention effect on reducing alcohol use in the 1 month following the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. engaged in regular heavy drinking, as indicated by consuming 5 or more drinks per occasion for men or 4 or more drinks per occasion for women at least 4 times in the month prior to enrollment
2. a score of ≥ 8 on the Alcohol Use Disorder Identification Test (AUDIT)

Exclusion Criteria:

1. under the age of 21
2. currently receiving treatment for alcohol problems, history of treatment in the 30 days before enrollment, or currently seeking treatment
3. a positive urine toxicology screen for any drug other than cannabis
4. a lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder
5. serious alcohol withdrawal symptoms
6. history of epilepsy, seizures, or severe head trauma
7. non-removable ferromagnetic objects in body
8. claustrophobia
9. pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Percent Heavy Drinking Days | 4 weeks post intervention
  Percent heavy drinking days defined as 5+ drinks for men and 4+ for women according to self-reported Timeline Follow Back (TLFB) data
Neural Alcohol Cue Reactivity | Single time point immediately post intervention
  Neural alcohol cue reactivity as measured by whole brain activation to alcohol taste cue vs. water taste cue using functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Lara A Ray, PhD, Principal Investigator — University of California, Los Angeles; Mitchell P Karno, PhD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grodin EN, Ray LA, MacKillop J, Lim AC, Karno MP. Elucidating the Effect of a Brief Drinking Intervention Using Neuroimaging: A Preliminary Study. Alcohol Clin Exp Res. 2019 Feb;43(2):367-377. doi: 10.1111/acer.13941. Epub 2019 Jan 20. PMID 30556913
- [Result] Grodin EN, Lim AC, MacKillop J, Karno MP, Ray LA. An Examination of Motivation to Change and Neural Alcohol Cue Reactivity Following a Brief Intervention. Front Psychiatry. 2019 Jun 11;10:408. doi: 10.3389/fpsyt.2019.00408. eCollection 2019. PMID 31244697
- [Derived] Meredith LR, Grodin EN, Karno MP, Montoya AK, MacKillop J, Lim AC, Ray LA. Preliminary study of alcohol problem severity and response to brief intervention. Addict Sci Clin Pract. 2021 Aug 24;16(1):54. doi: 10.1186/s13722-021-00262-6. PMID 34429151